CLINICAL TRIAL: NCT00947622
Title: Occipital Transcranial Direct Current Stimulation in Fibromyalgia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Prof. Dr. Dirk De Ridder, University Hospital Antwerp
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: TDCS_BP_FMS
Record Dates: First submitted 2009-07-27; First posted 2009-07-28 (Estimated); Last update posted 2009-07-28 (Estimated); Status verified 2009-07

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Neuromodulation; Transcranial Direct Current Stimulation; Occipital
MeSH Terms: conditions — Fibromyalgia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo stimulation (Placebo Comparator): Placebo stimulation at the occipital head area for 1800 seconds at 0 mA, three times a week, during one week (with seconds of stimulation to get onset tingling sensation)
  Interventions: Device: Transcranial direct current stimulation
- Effective transcranial stimulation (Experimental): Effective stimulation at the occipital head are for 1800 seconds at 2 mA, 3 times a week for 1 week
  Interventions: Device: Transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — Transcranial Direct current stimulation

SUMMARY:
The aim of this study is to investigate whether transcranial direct current stimulation is effective in the treatment of fibromyalgia related pain. The study provides a placebo arm and the design is a cross-over design.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from Fibromyalgia, diagnosed according to the criteria of the ACR-90, with exclusion of other pathologies mimicking the FMS related symptoms by a M.D. of the department of Physical Medicine and Rehabilitation (UZA, Belgium)
* Dutch speaking
* Stability of medication during the study

Exclusion Criteria:

* History of substance abuse, unless treated and in remission during 6 months
* Cardiac disease, implanted pace-maker or defibrillator
* History of epileptic insults
* Severe organic comorbidity
* Psychiatric comorbidity with psychotic symptoms
* Pregnancy

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2009-07; Primary Completion 2009-10 (Estimated); Study Completion 2009-11 (Estimated)

PRIMARY OUTCOMES:
Decrease on Visual Analogue Scale (VAS) score for Fibromyalgia related pain and pain scales of the Fibromyalgia Impact Questionnaire | baseline, directly after treatment, 3 weeks after treatment

SECONDARY OUTCOMES:
Changes in scores of the pain vigilance and awareness questionnaire, pain catastrophizing scale, fibromyalgia impact questionnaire and modified Fatigue Impact Scale | base line, directly after treatment and 3 weeks after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Dirk De Ridder, M.D. PhD., Study Chair — University Hospital, Antwerp; Mark Plazier, M.D., Principal Investigator — University Hospital, Antwerp
Locations (1):
- University Hospital Antwerp, Edegem, Antwerp, Belgium